CLINICAL TRIAL: NCT02508519
Title: Study of Zonal and Balance Acupuncture Pain Relief Effect
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Bogomolets National Medical University (Other)
Responsible Party: Principal Investigator, Golovchanskyi Oleksandr, M.D., Ph.D., Lecturer, Bogomolets National Medical University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: no grant number
Record Dates: First submitted 2015-07-21; First posted 2015-07-27 (Estimated); Last update posted 2015-08-17 (Estimated); Status verified 2015-08

CONDITIONS: Pain Syndrome
MeSH Terms: conditions — Somatoform Disorders | interventions — Acupuncture Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Zonal (Experimental): The zonal acupuncture group will receive a treatment according to a zonal method and a pain level will be estimated by the investigator according to a visual analog pain scale (VAS) before and 10 minutes and 15 minutes after the beginning of the treatment and the change of the pain level will be recorded. If possible the pain level will be measured again approximately 24 hours after the treatment and the change of the pain level will be again recorded.
  Interventions: Procedure: Acupuncture
- Balance (Experimental): The balance acupuncture group will receive a treatment according to a balance method, and a pain level will be estimated according to a visual analog pain scale (VAS) before and 10 minutes and 15 minutes after the beginning of the treatment and the change of the pain level will be recorded. If possible the pain level will be measured again approximately 24 hours after the treatment and the change of the pain level will be again recorded.
  Interventions: Procedure: Acupuncture
- Control (No Intervention): The control group will provide only the estimation of the the pain level according to a visual analog pain scale (VAS) but receive no acupuncture treatment. Then if possible the pain level will be measured again approximately 24 hours after the first measurement and the change of the pain level will be recorded.

INTERVENTIONS:
Procedure: Acupuncture — An acupuncture needle insertion according to zonal or balance method.
  Arms: Balance; Zonal

SUMMARY:
The aim of the study is to investigate how effective is zonal acupuncture method compared to balance method to obtain a short coming pain relief effect, which takes place several minutes after needle insertion.

DETAILED DESCRIPTION:
Main purpose of the study is to estimate the efficiency of the zonal acupuncture method compared to control group and the balance acupuncture method.

This study includes random completion of 3 groups of participants : zonal acupuncture, control group, balance acupuncture approximately 20 participants each.

The zonal acupuncture group will receive a treatment according to a zonal method and a pain level will be estimated by the investigator according to a visual analog pain scale (VAS) before and 10 minutes and 15 minutes after the beginning of the treatment and the change of the pain level will be recorded. If possible the pain level will be measured again approximately 24 hours after the treatment and the change of the pain level will be again recorded.

The control group will provide only the estimation of the the pain level according to a visual analog pain scale (VAS) but receive no acupuncture treatment. Then if possible the pain level will be measured again approximately 24 hours after the first measurement and the change of the pain level will be recorded for a control group too.

The balance acupuncture group will receive a treatment according to a balance method, and a pain level will be estimated according to a visual analog pain scale (VAS) before and 10 minutes and 15 minutes after the beginning of the treatment and the change of the pain level will be recorded. If possible the pain level will be measured again approximately 24 hours after the treatment and the change of the pain level will be again recorded.

These measurements are primary outcome of the experiment. Provided statistically consistent they will be treated to extract method efficiency estimation.

The participants from all tree groups may receive drug analgesia at some recorded moment of time before the procedure, however the investigators want to investigate the effect of acupuncture analgesia at the time when no other analgesia effect is present, so the investigators can exclude possible interference.

ELIGIBILITY:
Inclusion Criteria:

* post traumatic pain syndrome
* vertebrogenic pain syndrome

Exclusion Criteria:

* oncological diseases
* narcotic dependency
* psychiatric disorders

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2015-07; Primary Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Change of the Pain level on the VAS scale | 10 minutes, 15 minutes, 24 hours.
  Pain level is measured according to VAS scale before and 10 minutes and 15 minutes after the beginning of the treatment and the change of the pail level is recorded. If possible the pain level will be measured again approximately 24 hours after the treatment and the change of the pain level will be again recorded.